CLINICAL TRIAL: NCT02295696
Title: EMMA: Empowerment, Motivation and Medical Adherence
Acronym: EMMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Gitte Reventlov Husted, Researcher PhD, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: grhu
Record Dates: First submitted 2014-11-05; First posted 2014-11-20 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Adults, dialogue tools, outpatient clinic visits
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Intervention arm : EMMA consultations
  Interventions: Behavioral: EMMA
- Control group (No Intervention): Control arm: Usual care/consultations

INTERVENTIONS:
Behavioral: EMMA — Consultations using dialogue tools
  Arms: Intervention group

SUMMARY:
EMMA: Empowerment, Motivation and Medical Adherence. A consultation program based on dialogue tools for adults with poorly regulated Type 2 diabetes.

DETAILED DESCRIPTION:
Traditionally, the success of patients to manage their diabetes has been judged by their ability to adhere to a prescribed therapeutic regimen, and efforts have been spent developing strategies to promote adherence. It is estimated that 20% to 50% of patients with chronic conditions are not adherent to their prescribed medication regimen, with non-adherence being defined as <80% adherence to prescribed, relevant medication. The treatment regimen often comprises several elements such as poly-pharmacy including insulin administration, self-monitoring of blood glucose, diet and physical exercise. It is thus not just a matter of 'taking a pill or not' but implies lifestyle changes, knowledge and competence, and internal motivation for self-management. The investigators developed a consultation program based on dialogue tools. The EMMA program aims to support medication adherence and blood glucose control by facilitating rapport, exploring patient concerns and challenges, enabling knowledge exchange and supporting goal-setting and action-planning. A pilot test of the program appeared feasible and acceptable to patients and health care professionals and showed significant decrease on HbA1c. EMMA is now ready to be tested in a randomized controlled study (RCT) study.

ELIGIBILITY:
Inclusion Criteria:

* Adults Type 2 diabetes ≥ 18 år
* Type 2 diabetes ≥ 1 år
* HbA1c ≥ 64 mmol/mol (≥ 8%) at the last three measures before randomisation
* Taking medication for Type 2 diabetes • - Speak, read and understands Danish

Exclusion Criteria:

* Participating in other intervention research projects during the trial period
* Being treated by a psychiatrist or psychologist during the period
* Reduced sight or blindness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-08 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Baseline, 4½ month and 6 months after end of intervention period
  Change from baseline in HbA1c at 4½ month which is maintained or improved at 6 months

SECONDARY OUTCOMES:
Self-management | Baseline, 4½ month and 6 months after end of intervention period
  Change from baseline in Self-management skills at 4½ month assessed by increase in the Perceived Competence In Diabetes (PCD scale) which is maintained or improved at 6 months
Self-management | Baseline, 4½ month and 6 months after end of intervention period
  Change from baseline in Self-management skills at 4½ month assessed by increase in the Health Care Climate Questionnaire (HCCC scale) which is maintained or improved at 6 months
Self-management | Baseline, 4½ month and 6 months after end of intervention period
  Change from baseline in Self-management skills at 4½ month assessed by decrease in the Problem Areas in Diabetes Questionnaire (PAID scale) which is maintained or improved at 6 months
Self-management | Baseline, 4½ month and 6 months after end of intervention period
  Change from baseline in Self-management skills at 4½ month assessed by increase in The WHO5 Wellbeing Questionnaire (WHO5 scale) which is maintained or improved at 6 months
Self-management | Baseline, 4½ month and 6 months after end of intervention period
  Change from baseline in Self-management skills at 4½ month assessed by increase in the Treament Self-Regulation Questionnaire (TSRQ scale) which is maintained or improved at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gitte R Husted, PhD, Principal Investigator — Steno Diabetes Center, Denmark
Locations (1):
- Gitte R Husted, Gentofte Municipality, Denmark